CLINICAL TRIAL: NCT00661908
Title: Discrimination of Insulin-Treated Diabetic Subjects at the Workplace and by Insurances
Brief Title: Diabetes-Related Discrimination at Workplace and by Insurances
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Diabetes Association Basel (Other)
Responsible Party: Piera M Nebiker, MD, University Hospital of Basel, Switzerland
Other Study IDs: 274/03
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Insulin-Treated Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: insulin-treated diabetic subjects of North-western part of Switzerland

SUMMARY:
Diabetic subjects often report of problems at the workplace or when contracting insurances because of their diabetes.

By distributing a self-report questionnaire to insulin-treated Type 1 and Type 2 diabetic subjects we wanted to analyse the frequency of work- and insurance-related discrimination. Furthermore we wanted to detect socio-demographic and diabetes-related factors which are associated with increased discrimination at workplace and by insurances. We hypothesized that diabetes-related discrimination at workplace and by insurances exists and that certain factors like having severe hypoglycaemic events, being type 1 diabetic or being overweight would be associated with more problems at work or with insurances.

DETAILED DESCRIPTION:
Our self report questionnaire included 83 items to assess treatment goals, quality of life and discrimination at workplace or by insurances. 636 questionnaires were distributed and were answered and returned. Anonymity was ensured. Patients were recruited from the diabetes outpatient clinic of the University of Basel Hospital, 5 regional hospitals, specialist practices and general practitioner practices.

The aims of this study are to investigate the prevalence of discrimination at workplace and by insurances due to diabetes mellitus. Furthermore we want analyse if socio-demographic factors (age,gender,origin) show an impact on diabetes-related discrimination at workplace and by insurances. We hypothesize furthermore that certain diabetes-related factors like having severe hypoglycemias, being type 1 diabetic, having diabetic complications or being overweight/obese is associated with more problems at work and with insurances.

Data will be analysed by a multiple ordinal regression analysis. We will correct data for age, gender, employment status and diabetes type.

ELIGIBILITY:
Inclusion Criteria:

* german-speaking insulin-treated diabetic patients

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Within a time period of two month we recruited all insulin-treated diabetic patients from the outpatient clinic of the University Hospital of Basel (n=203), from 5 regional hospitals (n=135) in the North-western part of Switzerland and from 13 specialist practices (n=107) as well as from 15 randomly selected general practioner practices (n=64)in the mentioned area.
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2004-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piera M Nebiker, MD, Principal Investigator — University of Basel